CLINICAL TRIAL: NCT02078687
Title: Growth, Risks of Allergy and Metabolic Syndrome in 6 Year Old Children Born Preterm Compared to Nutrition in the First Four Month After Hospital Discharge
Brief Title: Growth, Risks of Allergy and Metabolic Syndrome in 6 Year Old Children Born Preterm Compared to Postdischarge Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Holbaek Sygehus (Other); Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Line Toftlund, PhD student, doctor in medicine, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDU-2014-LHT
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Infant, Very Low Birth Weight; Metabolic Syndrome, Protection Against; Allergy; Dietary Modification
Keywords: very preterm; nutrition; 6 year follow-up; growth; metabolic syndrome; allergy; dexa
MeSH Terms: conditions — Metabolic Syndrome; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1, HM (Active Comparator): This group received breastfeeding (human milk, HM) solely throughout the 4 month of intervention. Randomisation for group 1 or group 2. Mothers own milk.
  Interventions: Dietary Supplement: Mothers own milk
- Group 2, HMF (Active Comparator): This group received mothers own milk with fortification (human milk fortification, HMF) throughout the 4 month intervention period. Randomisation for group 1 og group 2. Enfamil HM fortifier, Mead Johnson.
  Interventions: Dietary Supplement: Enfamil HM fortifier, Mead Johnson; Dietary Supplement: Mothers own milk
- Group 3, PF (Active Comparator): This group received preterm formula (PF) throughout the intervention period of 4 month. This group was not randomised for ethical reasons. Enfalac Premature Formula, Mead Johnson Nutritionals
  Interventions: Dietary Supplement: Enfalac Premature Formula, Mead Johnson Nutritionals

INTERVENTIONS:
Dietary Supplement: Enfamil HM fortifier, Mead Johnson — Enfamil was added to a small amount of mothers expressed milk and given in a bottle or with a small cup every day. Group 2 (HMF) received 5 packets each day for 4 month containing; 17.5 kcal, 1.375 g protein/ 5 packets
  Other Names: Enfamil HM fortifier, Mead Johnson, Njimegen, Netherlands
  Arms: Group 2, HMF
Dietary Supplement: Enfalac Premature Formula, Mead Johnson Nutritionals — Group 3 received Enfalac containing:
  68 kcal, 2 g protein, 7.4 g carbohydrate, 3.5 g fat/ 100 ml
  Other Names: Enfalac PF, Mead Johnson Nutritionals, Njimegen, Netherlands
  Arms: Group 3, PF
Dietary Supplement: Mothers own milk — Group 1 received mothers own milk without fortification
  Arms: Group 1, HM; Group 2, HMF

SUMMARY:
This is a follow-up cohort study of 6 years old children born preterm in Denmark from 2004-2008, and at four different neonatal units. During hospitalisation they received breast milk with fortification. At time of discharge there were made 3 different nutrition groups; if possible they were randomised into one of two groups:

1. Breastfeeding solely
2. Breastfeeding with fortification

   If breastfeeding was not possible they were put in group 3 and were bottle fed with:
3. Preterm formula

This nutrition intervention went on for 4 month. At the age of 6, the children will be invited to come for an ambulant control and other examinations regarding growth, allergy and metabolic syndrome.

DETAILED DESCRIPTION:
Project background:

The study is based on a follow-up of a cohort of very preterm infants born before week 32, as at discharge from the neonatal departments were randomized to a protein supplement or not while breastfeeding after discharge. If the preterm child was not breastfed, it received a premature infant formula after discharge. Since we have three groups of prematures, which are fed differently after discharge, it is useful to follow up at 6 years of age and specifically examine the following areas:

Metabolic syndrome:

Unlike the past, the survival rate of very preterm infants is now high. Most is expected to survive. The question is the extent to which these children have increased morbidity compared with children born at term, and their quality of life is affected by the fact that they are born prematurely. There has previously been shown a link between children born SGA and later development of type 2 diabetes mellitus, hypertension, ischemic heart disease and cerebrovascular disasters. Too rapid catch-up growth also increases the possible risk of developing metabolic syndrome in the mature child. The question is whether this is also the case in children born prematurely and whether the risk is the same. The problem is just that you want to provide them with adequate amino acids for protein synthesis, as they approach the growth of peers fetuses and also ensure the development of the brain with essential fatty acids, but maybe they can not tolerate a too rapid "catch-up" - growth.

A study comparing preterm born children aged 4-10 years with mature children born of the same age found that the group with preterm births had increased systolic and diastolic blood pressure and higher insulin levels. This was true regardless of whether the children were born SGA and AGA at birth. This concluded that there were metabolic abnormalities in preterm similar to those found in children born at term but SGA. The same article mentions the concept of "fetal programming". This covers a hypothesis which suggests that a fetus at risk in the uterus will adapt best to survive, and this adjustment will be permanent.

The same team has published an article, which have found impaired insulin sensitivity in preterm infants (SGA and AGA) compared to mature AGA children. Insulin sensitivity is greatest in the mature AGA. Next comes the mature SGA and eventually the premature. To show the importance of this area, they point out that out of those who have diabetes mellitus type 2, 35% has had low birth weight.

In trying to find a way it will be interesting, and very relevant, to see if diet the first months of life have an impact on these metabolic complications later in life.

Allergy:

It is unknown whether preterms are at increased risk of developing allergic symptoms. Breastfeeding reduces the risk of developing allergic diseases, while cow milk-based infant formulas increase the risk. The preterm infants in this study completed during hospitalization with fortifier containing cow's milk protein, and the preterm infant formula is cow milk based. It is therefore interesting to see if there is an increased incidence of allergic symptoms in one of the groups. An article formed on the basis of a study of two groups of children, one group consisted of children with a birth weight less than 1500 g, and the second group consisted of children with a birth weight over 2500 g, describes that there was no difference in the incidence of atopy. Another study studied the incidence of food allergies in an area of 13,980 children, and found that 4.23 % were diagnosed with this at the age of six. There was no difference in the incidence of categorization in GA.

The first study mentioned above studied also the appearance of wheezing. This was done using spirometry. The result was that the lifetime risk of preterm births was 43% for developing wheezing, while it was only 17% in mature births. Besides wheezing low GA at birth was associated with decreased lung capacity, reduced forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) and asthma. A relevant question is whether children develop these respiratory symptoms solely on the basis that they are born preterm or nutritional type influences the risk of its development.

Growth and catch-up:

Some studies have gradually studied prematurely born children's growth compared to some control children - especially in the first period after discharge from the neonatal units. As we know, human milk has the best composition in relation to children's needs. There has been made a study on nutrition of preterms with human milk against fortified human milk which states that those who get pure milk, are at greatest risk of malnutrition by discharge and that it is a good strategy to provide breast milk multinutrient enrichment. In the study mothers milked out half of their daily quantity for enrichment. Though, they request long-term studies to determine the long-term effects of it.

Other studies have followed prematurely born children up to 20 years of age and 11 years of age and were compared with a control group of normal weight, not preterm births. Outcome was height, weight, BMI. In one case also head circumference. One study concludes that all very low birthweight children (VLBW) were smaller than the control group. In particular SGA boys were smaller. The second study concluded that extremely immature children have poor growth in early childhood, but they have catch-up until 11 years of age. All prematures remain less than the control group.

A comparison of both nutrition after discharge and follow-up beyond 1 year of age will be very interesting to be able to optimize nutrition and growth of extremely premature infants, both AGA and SGA.

A dual-energy X-ray absorptiometry (DEXA) scan is a study that reveals body composition of bone, muscle and fat. A study of whether the scanning can be used to detect body composition, concluded that DEXA is a good tool for this. It is a quick (minutes) survey that provides minimal radiation, and it is interesting because a scan of the 3 groups in this project will elucidate whether there is a difference in body composition and thus whether a nutritional type provides better basis for the best growth. The same study, which was built on an RCT (randomized controlled trial) of 33 children with GA less than 35 weeks and a birth weight below 1,750 grams who received either 1) standard replacement or 2) enriched compensation for 2 months after discharge, found no difference in body composition or weight gain. It calls for larger studies with longer follow-up. Another study, just as this PhD project, divide the children into several groups depending on Nutrition (1: enriched substitute 2: standard replacement 3: human breast milk), found by DEXA scanning at 6 months of age, group 1 had lower fat mass and group 3 had lower lean (muscle) mass and higher fat mass. So, there is a difference in body composition depending on nutrition. It may sound logical, but will it affect children later in life? - and if so, in what way? From the above examples of previous studies, one can conclude that the optimal nutrition of preterms is under development and there is a continued lack of clarification of how preterm infants grow after discharge and whether one type of nutrition is better.

Hypotheses:

* Nutrition after discharge does affect premature children's growth in the first years of life.
* Catch-up growth proceeds after 1 year of age.
* The growth pattern for prematures born SGA is different from prematures born AGA.
* There is no increase in allergies between prematures, who was fed with premature formula or enriched mothers milk before and after discharge compared with mothers milk without enrichment.
* Premature children fed with a preterm formula have an extended risk for developing metabolic syndrome on basis of excessive growth the first months of life.
* It is possible that premature SGA children have greater risks of developing metabolic syndrome on the basis of excessive growth the first month of life.
* Fat mass and lean mass vary among prematures depending on the nutrition the first month after discharge.

Purpose of the project:

1. Investigate whether there are long-term effect on growth after cessation of enrichment of breast milk in 2, 3 and 6 years of age.
2. Examine the relationship between protein intake to 4 months of age (corrected) and blood pressure, HbA1c and serum cholesterol by 6 years of age.
3. Uncover the incidence of allergy symptoms from the eyes and nose, skin, stomach / intestinal and respiratory tract incl affected lung function in children born prematurely.
4. Elucidate whether there is an increased risk of metabolic syndrome in children born prematurely and nourished in different ways.
5. Investigate whether preterms have different fat distribution and nutrition up to 4 months corrected age affect them.
6. Illuminate catch-up growth in children born prematurely and up to 6 years of age.

Planned studies:

1. Weight, height, head circumference, blood pressure
2. Registration of any allergy symptoms and airway symptoms.
3. Blood tests for diabetes, screening for metabolic syndrome and allergies.
4. Questionaires to investigate allergy symptoms.
5. A dexa scan to see the body composition of fat, muscle and bone.

Randomization:

The children were randomized when they could eat (breast or bottle) at gestational age 34-42. Twins and triplets were randomly assigned to the same group.

At randomization an impartial person in the department the child was hospitalized in, pulled an envelope with information on what kind of nutrition, the child should have after discharge and up to 4 months of corrected age.

Statistics:

Originally, there were strength calculations prior to randomization in the project. This showed that there were needed 85 children in each feeding group. A total of 320 children in the original project were enrolled. However, there has been a waiver until 1 year of age, and there are 278 children remaining to follow-up.

Wilcoxon rank-sum test or t-test for continuous variables, and if categorical variables chi2test will be used to compare the nutritional groups.

Multiple logistic regression models will be used to compare the clinical relevant variables that have possible influence on the growth of various dietary groups.

Growth will be analyzed from Z-score and delta z-score and will be calculated from a relevant reference for comparing nutritional groups growth.

Allergy risks and metabolic syndrome will be calculated using the above methods and odds ratio.

Project Period:

From 2004 - 2008 there were formed three groups of preterm children at clinical randomization. A Ph.D. dissertation was made subsequently dealing with preterm growth up to 1 year of age, nutrition and composition of breast milk of mothers of preterm babies.

Between the ages of 2 and 3 years, children have come to control for a follow-up Ph.D. The children become 6 years from July 2010 - 2014, where they also will be invited to a follow-up check on the current Ph.D. project.

The children will be followed up in their respective departments / hospitals in Kolding, Skejby, Holbæk and Odense.

Ethical considerations:

For inclusion in the randomized controlled study parents signed an acceptance which included follow-up at 6 years of age.

The initial randomized controlled study was approved by the Ethics Committee 1 July 2004 (J. Nr.VF20030208). As part of the 6-year follow-up, there is added and approved Protocol 1-8.

In addition, permission from the Data Inspectorate of the original project with change in 2007 (J. No 2007-41-1349) is extended until 2016.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the original study when they were discharge from hospital
* Parents accept of participation in the 6 year follow-up

Exclusion Criteria:

* Participation not accepted by parents
* Genetic diseases with influence on growth

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Growth | Follow-up at approximately 6 years corrected age
  Measurement of weight at 6 years corrected age

SECONDARY OUTCOMES:
Metabolic syndrome | Follow-up at approximately 6 years corrected age
  Dexa scan including fat mass, muscle mass, bone mass and Body Mass Index.

OTHER OUTCOMES:
Allergy | Follow-up at approximately 6 years corrected age
  Test for lung function: body box breathing test
Growth | Follow-up at approximately 6 years corrected age
  Lenght at 6 years corrected age
Growth | Follow-up at approximately 6 years corrected age
  Head circumference at 6 years corrected age
Metabolic syndrome | Follow-up at approximately 6 years corrected age
  Blood test; blood glucose, HbA1c, HDL, insulin, Insulin-like growth factor 1 (IgF1), C-peptide
Metabolic syndrome | Follow-up at approximately 6 years corrected age
  Blood pressure
Allergy | Follow-up at approximately 6 years corrected age
  Allergy questionnaire
Allergy | Follow-up at approximately 6 years corrected age
  blood samples; Immunoglobulin E (IgE)
Allergy | Follow-up at approximately 6 years corrected age
  Lung function: NO-test

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Zachariassen, Specialist, Study Director — HC Anderson Children´s Hospital, OUH, Denmark; Susanne Halken, Professor, Study Chair — HC Anderson children´s Hospital, OUH, Denmark; Lone Agertoft, Specialist, Study Director — HC Anderson children´s Hospital, OUH, Denmark; Line H Toftlund, MD, Principal Investigator — HC Anderson children´s Hospital, OUH, Denmark
Locations (1):
- HC Anderson Children´s Hospital, OUH, Odense, Denmark

REFERENCES:
- [Background] Barker DJ. In utero programming of chronic disease. Clin Sci (Lond). 1998 Aug;95(2):115-28. PMID 9680492
- [Background] Hofman PL, Regan F, Harris M, Robinson E, Jackson W, Cutfield WS. The metabolic consequences of prematurity. Growth Horm IGF Res. 2004 Jun;14 Suppl A:S136-9. doi: 10.1016/j.ghir.2004.03.029. PMID 15135796
- [Background] Amesz EM, Schaafsma A, Cranendonk A, Lafeber HN. Optimal growth and lower fat mass in preterm infants fed a protein-enriched postdischarge formula. J Pediatr Gastroenterol Nutr. 2010 Feb;50(2):200-7. doi: 10.1097/MPG.0b013e3181a8150d. PMID 19881394
- [Background] Hofman PL, Regan F, Jackson WE, Jefferies C, Knight DB, Robinson EM, Cutfield WS. Premature birth and later insulin resistance. N Engl J Med. 2004 Nov 18;351(21):2179-86. doi: 10.1056/NEJMoa042275. PMID 15548778
- [Background] Siltanen M, Savilahti E, Pohjavuori M, Kajosaari M. Respiratory symptoms and lung function in relation to atopy in children born preterm. Pediatr Pulmonol. 2004 Jan;37(1):43-9. doi: 10.1002/ppul.10402. PMID 14679488
- [Background] Liem JJ, Kozyrskyj AL, Huq SI, Becker AB. The risk of developing food allergy in premature or low-birth-weight children. J Allergy Clin Immunol. 2007 May;119(5):1203-9. doi: 10.1016/j.jaci.2006.12.671. Epub 2007 Mar 26. PMID 17379288
- [Background] G. Zachariassen, J Færk mf. Nutrient-enrichment of human milk for preterm infants after hospital discharge - a randomized controlled trial. Pediatrics 2010.
- [Background] O'Connor DL, Khan S, Weishuhn K, Vaughan J, Jefferies A, Campbell DM, Asztalos E, Feldman M, Rovet J, Westall C, Whyte H; Postdischarge Feeding Study Group. Growth and nutrient intakes of human milk-fed preterm infants provided with extra energy and nutrients after hospital discharge. Pediatrics. 2008 Apr;121(4):766-76. doi: 10.1542/peds.2007-0054. PMID 18381542
- [Background] Hack M, Schluchter M, Cartar L, Rahman M, Cuttler L, Borawski E. Growth of very low birth weight infants to age 20 years. Pediatrics. 2003 Jul;112(1 Pt 1):e30-8. doi: 10.1542/peds.112.1.e30. PMID 12837903
- [Background] Farooqi A, Hagglof B, Sedin G, Gothefors L, Serenius F. Growth in 10- to 12-year-old children born at 23 to 25 weeks' gestation in the 1990s: a Swedish national prospective follow-up study. Pediatrics. 2006 Nov;118(5):e1452-65. doi: 10.1542/peds.2006-1069. PMID 17079546
- [Background] De Curtis M, Pieltain C, Rigo J. Body composition in preterm infants fed standard term or enriched formula after hospital discharge. Eur J Nutr. 2002 Aug;41(4):177-82. doi: 10.1007/s00394-002-0374-2. PMID 12242586
- [Background] Zachariassen G, Faerk J, Grytter C, Esberg BH, Hjelmborg J, Mortensen S, Thybo Christesen H, Halken S. Nutrient enrichment of mother's milk and growth of very preterm infants after hospital discharge. Pediatrics. 2011 Apr;127(4):e995-e1003. doi: 10.1542/peds.2010-0723. Epub 2011 Mar 14. PMID 21402642
- [Background] Zachariassen G, Faerk J, Esberg BH, Fenger-Gron J, Mortensen S, Christesen HT, Halken S. Allergic diseases among very preterm infants according to nutrition after hospital discharge. Pediatr Allergy Immunol. 2011 Aug;22(5):515-20. doi: 10.1111/j.1399-3038.2010.01102.x. Epub 2011 Feb 20. PMID 21332800
- [Derived] Toftlund LH, Halken S, Agertoft L, Zachariassen G. Early nutrition and signs of metabolic syndrome at 6 y of age in children born very preterm. Am J Clin Nutr. 2018 May 1;107(5):717-724. doi: 10.1093/ajcn/nqy015. PMID 29722837